CLINICAL TRIAL: NCT00191451
Title: Phase II Trial of Gemzar Plus Paraplatin (Plus Herceptin in HER2+ Patients) in Metastatic Breast Cancer
Brief Title: A Study of Gemcitabine and Carboplatin (Plus Herceptin in Human Epidermal Growth Factor Receptor 2 Positive [HER2+] Patients) With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9397; B9E-US-S359
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Carboplatin; Trastuzumab

ARMS (3):
- HER2+ (Experimental): Human Epidermal growth factor Receptor 2 positive (HER2+): Gemcitabine + Carboplatin + Herceptin.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Herceptin
- HER2- (Taxane-) (Experimental): Human Epidermal growth factor Receptor 2 negative (HER2-): Gemcitabine + Carboplatin. (Taxane-naive patients).
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- HER2- (Taxane+) (Experimental): Human Epidermal growth factor Receptor 2 negative (HER2-): Gemcitabine + Carboplatin. (Taxane-pretreated patients).
  Interventions: Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine — Day 1 of 14 day cycle (Cycles 1-9):1500 milligram per square meter (mg/m2) intravenous (IV) (30 minute infusion)
  Other Names: Gemzar
Drug: Carboplatin — Day 1 of 14 day cycle (Cycles 1-9): Carboplatin area under the curve (AUC)=2.5 intravenous (IV) (30-60 minute infusion).
  Other Names: Paraplatin
Drug: Herceptin — Day 1 of 14 day cycle (Cycle 1): 8 milligrams per kilogram (mg/kg) intravenous (IV) (90 minute infusion).
  Day 1 of 14 day cycle (Cycles 2-9): 4 mg/kg IV (30 minute infusion). Day 1 of 21 day cycle (Cycles 10+): 6 mg/kg IV (30 minute infusion).
  Arms: HER2+

SUMMARY:
The purposes of this study are to determine the safety of gemcitabine and paraplatin either with or without trastuzumab Any side effects that might be associated with these compounds. Whether the two or three drugs listed above when given in combination can help patients with metastatic breast cancer. How long the treatment will stop the growth of the cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of metastatic breast cancer
2. Able to visit the doctor's office at least every 14 days during the actual treatment
3. Able to care for yourself, even if you cannot work or participate in other normal activities
4. Your blood results must be adequate for therapy.
5. If you are a female of childbearing potential and test negative for pregnancy, use a reliable method of birth control during and for three months following the last dose of study drug.

Exclusion Criteria:

1. Have received gemcitabine, paraplatin, or trastuzumab for your cancer.
2. Be pregnant or breastfeeding
3. Have cancer to the brain and has not been treated
4. Have another active cancer besides breast cancer
5. Have received stem cell or bone marrow transplant for hematologic (blood type) cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-04; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HER2+: Human Epidermal growth factor Receptor 2 positive: Gemcitabine + Carboplatin + Herceptin.
  Gemcitabine: Day 1 of 14 day cycle (Cycles 1-9):1500 milligram per square meter (mg/m2) intravenous (IV) (30 minute infusion); Carboplatin: Day 1 of 14 day cycle (Cycles 1-9): Carboplatin area under the curve (AUC)=2.5 intravenous (IV) (30-60 minute infusion); Herceptin: Day 1 of 14 day cycle (Cycle 1): 8 milligrams per kilogram (mg/kg) intravenous (IV) (90 minute infusion). Day 1 of 14 day cycle (Cycles 2-9): 4 mg/kg IV (30 minute infusion). Day 1 of 21 day cycle (Cycles 10+): 6 mg/kg IV (30 minute infusion).
- HER2- (Taxane-): Human Epidermal growth factor Receptor 2 negative: Gemcitabine + Carboplatin. (Taxane-naive patients).
  Gemcitabine: Day 1 of 14 day cycle (Cycles 1-9):1500 milligram per square meter (mg/m2) intravenous (IV) (30 minute infusion); Carboplatin: Day 1 of 14 day cycle (Cycles 1-9): Carboplatin area under the curve (AUC)=2.5 intravenous (IV) (30-60 minute infusion).
- HER2- (Taxane+): Human Epidermal growth factor Receptor 2 negative: Gemcitabine + Carboplatin. (Taxane-pretreated patients).
  Gemcitabine: Day 1 of 14 day cycle (Cycles 1-9):1500 milligram per square meter (mg/m2) intravenous (IV) (30 minute infusion); Carboplatin: Day 1 of 14 day cycle (Cycles 1-9): Carboplatin area under the curve (AUC)=2.5 intravenous (IV) (30-60 minute infusion).
Period: Overall Study
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Started | 50 | 51 | 49
Received at Least One Dose of Study Drug | 50 | 48 | 47
Completed | 43 | 37 | 35
Not Completed | 7 | 14 | 14
Not completed — Withdrawal by Subject | 2 | 3 | 5
Not completed — Physician Decision | 2 | 9 | 6
Not completed — Sponsor Decision | 1 | 0 | 0
Not completed — Ineligible | 0 | 1 | 0
Not completed — Reason Not Specified | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+) | Total
Number analyzed (Participants) | 50 | 51 | 49 | 150
Age Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.45) | 55.7 (11.17) | 54.8 (9.92) | 55.55 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 49 | 150
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 49 | 150
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (Fully Active) to 5 (Death).
  participants
    0 - Fully Active | 41 | 36 | 32 | 109
    1 - Ambulatory, Restricted Strenuous Activity | 8 | 14 | 17 | 39
    2 - Ambulatory, No Work Activities | 1 | 1 | 0 | 2
Race/Ethnicity [Number; unit: participants]
  Caucasian | 31 | 42 | 36 | 109
  Black | 8 | 5 | 11 | 24
  Hispanic | 7 | 4 | 1 | 12
  Other | 4 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response=30% decrease in sum of longest diameter of target lesions; Progressive Disease=20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria.
Time Frame: baseline to disease progression/recurrence (up to 3.5 years)
Population: Efficacy evaluable subjects include all subjects who received at least 2 cycles of treatment with at least 1 follow-up tumor assessment, and did not violate the protocol in any fundamental manner related to the evaluation of efficacy.
Measure: Number; unit: participants
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Number analyzed (Participants) | 50 | 47 | 47
participants
  Complete Response (CR) | 6 | 0 | 1
  Partial Response (PR) | 26 | 13 | 15
  Stable Disease (SD) | 12 | 20 | 13
  Progressive Disease (PD) | 4 | 12 | 17
  Not Evaluable (NE) | 2 | 2 | 1

2. Secondary Outcome: Duration of Response
Description: Among tumor responders, the duration of tumor response is measured from the date of response (complete response [CR] or partial response [PR]) until the first date of documented progression or death from any cause. Duration of tumor response will be censored at the date of the last follow-up visit for tumor responders who are still alive and who have not progressed.
Time Frame: date of response (CR or PR) until the first date of documented progression or death from any cause (up to 3.5 years)
Population: Number of patients with complete or partial response. Censored patients: 6 in HER2+, 6 in HER2- (Taxane-), and 5 in HER2- (Taxane+).
Measure: Median (Full Range); unit: months
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Number analyzed (Participants) | 32 | 13 | 16
months | 6.9 [2.0 to 42.1] | 6.4 [3.5 to 29.7] | 5.6 [2.3 to 14.8]

3. Secondary Outcome: Number of Patients Who Experienced Alopecia
Time Frame: Baseline to 3.5 years
Population: Number of patients who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Number analyzed (Participants) | 50 | 48 | 47
participants | 21 | 17 | 16

4. Secondary Outcome: Time to Disease Progression (TTP)
Description: If a patient is lost to follow-up, the patient will be censored as of the last date of contact. Patients who start a new treatment before they progress will be censored as of the date of start of the new treatment. If a patient died due to reason other than study disease, and patient has not progressed or received any new treatment, TTP is censored at the date of death.
Time Frame: randomization date to the earliest date of the first documented disease progression date or the date of death if the patient dies due to study disease (up to 3.5 years)
Population: Intent to treat population: all randomized patients. Censored patients: 10 in HER2+, 20 in HER2- (Taxane-), and 12 in HER2- (Taxane+).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Number analyzed (Participants) | 50 | 51 | 49
months | 7.2 [6.0 to 9.0] | 5.6 [3.3 to 7.2] | 4.6 [1.8 to 9.0]

5. Secondary Outcome: Percentage of Patients With Overall Survival at 1 Year and 2 Years
Description: Kaplan-Meier estimates of overall survival (percentage of patients surviving) at 1 year and 2 years.
Time Frame: 1 Year, 2 Years
Population: Intent to treat population: all randomized patients. Censored patients: 31 HER2+; 19 HER2- (Taxane-); 9 HER2- (Taxane+).
Measure: Number; unit: percentage of participants
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Number analyzed (Participants) | 50 | 51 | 49
percentage of participants
  1 Year Overall Survival | 90.0 | 67.5 | 47.8
  2 Year Overall Survival | 73.3 | 41.4 | 20.5

ADVERSE EVENTS:
Description: Adverse events are provided for all patients who received at least one dose of study drug. Adverse events represent all grades (I-IV).
Arm/Group | HER2+ | HER2- (Taxane-) | HER2- (Taxane+)
Serious Adverse Events (participants affected / at risk) | 10/50 | 11/48 | 10/47
Other Adverse Events (participants affected / at risk) | 50/50 | 48/48 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2+ (N=50) | HER2- (Taxane-) (N=48) | HER2- (Taxane+) (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mucous membrane disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (5) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HER2+ (N=50) | HER2- (Taxane-) (N=48) | HER2- (Taxane+) (N=47)
Anaemia (Blood and lymphatic system disorders) | 31 (60) | 24 (35) | 22 (35)
Leukopenia (Blood and lymphatic system disorders) | 16 (47) | 20 (64) | 10 (29)
Lymphopenia (Blood and lymphatic system disorders) | 4 (11) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 35 (102) | 37 (109) | 28 (77)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (34) | 17 (47) | 15 (32)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 5 (7) | 0 (0)
Lacrimation increased (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 19 (27) | 19 (30) | 14 (18)
Diarrhoea (Gastrointestinal disorders) | 10 (17) | 13 (20) | 8 (9)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 27 (59) | 33 (71) | 22 (44)
Stomatitis (Gastrointestinal disorders) | 7 (8) | 6 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (17) | 18 (32) | 12 (21)
Asthenia (General disorders) | 1 (1) | 6 (8) | 3 (4)
Chest discomfort (General disorders) | 3 (3) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (5) | 5 (5) | 6 (6)
Chills (General disorders) | 4 (5) | 7 (9) | 5 (6)
Fatigue (General disorders) | 37 (70) | 35 (56) | 30 (50)
Mucosal inflammation (General disorders) | 1 (2) | 3 (4) | 4 (4)
Oedema (General disorders) | 4 (5) | 5 (5) | 2 (2)
Oedema peripheral (General disorders) | 5 (7) | 6 (8) | 10 (11)
Pain (General disorders) | 3 (3) | 2 (2) | 6 (6)
Pyrexia (General disorders) | 6 (7) | 4 (5) | 5 (8)
Rhinitis (Infections and infestations) | 6 (6) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 3 (3)
Alanine aminotransferase (Investigations) | 6 (8) | 7 (7) | 1 (2)
Alanine aminotransferase increased (Investigations) | 10 (16) | 10 (14) | 7 (8)
Aspartate aminotransferase (Investigations) | 4 (5) | 5 (6) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 10 (16) | 12 (16) | 5 (7)
Blood alkaline phosphatase (Investigations) | 3 (3) | 0 (0) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 8 (10) | 5 (5) | 5 (6)
Blood calcium decreased (Investigations) | 2 (2) | 3 (3) | 1 (3)
Blood glucose increased (Investigations) | 2 (4) | 3 (5) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Haemoglobin (Investigations) | 11 (11) | 9 (10) | 7 (9)
Haemoglobin decreased (Investigations) | 2 (6) | 7 (11) | 2 (3)
Neutrophil count (Investigations) | 5 (10) | 2 (2) | 1 (3)
Platelet count (Investigations) | 4 (11) | 8 (16) | 7 (12)
Platelet count increased (Investigations) | 3 (3) | 0 (0) | 0 (0)
White blood cell count (Investigations) | 6 (15) | 5 (10) | 8 (15)
White blood cell count decreased (Investigations) | 3 (9) | 2 (2) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 8 (11) | 11 (13) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 3 (5) | 4 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (23) | 8 (13) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (7) | 4 (6) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 9 (16) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 5 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (19) | 6 (12) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (9) | 5 (5)
Dizziness (Nervous system disorders) | 4 (6) | 10 (15) | 4 (4)
Dysgeusia (Nervous system disorders) | 5 (10) | 7 (9) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 2 (2) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 4 (6) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (5) | 4 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 7 (7) | 4 (5) | 8 (8)
Depression (Psychiatric disorders) | 3 (3) | 3 (3) | 7 (7)
Insomnia (Psychiatric disorders) | 9 (9) | 11 (12) | 4 (4)
Breast pain (Reproductive system and breast disorders) | 3 (3) | 2 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (24) | 11 (14) | 10 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 7 (10) | 11 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 21 (22) | 17 (22) | 16 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 3 (5) | 4 (5)
Rash (Skin and subcutaneous tissue disorders) | 11 (14) | 7 (9) | 5 (5)
Hot flush (Vascular disorders) | 4 (5) | 7 (8) | 4 (4)
Lymphoedema (Vascular disorders) | 1 (1) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days